CLINICAL TRIAL: NCT05777837
Title: Laparoscopic Excision Versus Combined Hysteroscopic and Laparoscopic Repair Without Excision of Large Cesarean Scar Niche: A Randomized Controlled Trial
Brief Title: Laparoscopic Versus Combined Laparoscopic and Hysteroscopic Repair of CS Niche
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mahmoud Abubakr Negm, lecturer of Obstetrics and gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS scar niche repair
Record Dates: First submitted 2023-02-25; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Scar Niche

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Excision of Large Cesarean Scar Niche (Active Comparator)
  Interventions: Procedure: laparoscopic repair of cesarean scar niche
- Combined Hysteroscopic and Laparoscopic Repair without Excision of Large Cesarean Scar Niche (Active Comparator)
  Interventions: Procedure: Combined hysteroscopic and laparoscopic repair of cesarean scar niche

INTERVENTIONS:
Procedure: laparoscopic repair of cesarean scar niche — Intentional perforation of the niche will be done using uterine sound and excision of the fibrotic edges then suturing the uterine incision using 2-0 absorbable suture.
  Other Names: laparoscopic excision of cesarean scar niche
  Arms: Laparoscopic Excision of Large Cesarean Scar Niche
Procedure: Combined hysteroscopic and laparoscopic repair of cesarean scar niche — Hysteroscopic resection of the niche under laparoscopic guide will be done to avoid perforation of the niche. After completion of the hysteroscopic approach, laparoscopic plication of the niche without opening it will be done using multiple interrupted 2-0 absorbable suture.
  Other Names: Combined hysteroscopic and laparoscopic repair without excision of large cesarean scar niche
  Arms: Combined Hysteroscopic and Laparoscopic Repair without Excision of Large Cesarean Scar Niche

SUMMARY:
Uterine niche is a frequent condition in patients with a history of cesarean section. Many treatment methods have been described for repair of niche with varying effectivities. In conventional Laparoscopic approach, not all bleeding points and fibrotic area are resected, while conventional hysteroscopic one result in more wide defect with high risk of recurrence and cannot be used in large niche with low RMT. In this new Double approach (hysteroscopy and laparoscopy) technique, the benefit of both laparoscopy and hysteroscopy will be attained.

DETAILED DESCRIPTION:
In all patient involved in the study, laparoscopic entry will be done, then adhesiolysis and creation of the bladder flap(dissection of the bladder from the uterine scar) then:

Group (I): Laparoscopic Excision of large cesarean scar niche:

Intentional perforation of the niche will be done using uterine sound and excision of the fibrotic edges then suturing the uterine incision using 2-0 absorbable suture.

Group (II): Combined hysteroscopic and laparoscopic repair without excision of large cesarean scar niche:

The investigators will do the hysteroscopic resection of the niche under laparoscopic guide to avoid perforation of the niche. After completion of the hysteroscopic approach, laparoscopic plication of the niche without opening it will be done using multiple interrupted 2-0 absorbable suture After suturing, the hysteroscopy will be introduced again to assess the repair The patient will be sent home the day after. They will be followed up after 3 and 6 months.

Checkup of CSD repair:

After 6 month of surgery both groups will be examined using sonohysterography to assess the changes in niche diameters

Core outcome sets:

* Enlargement of the residual myometrium thickness and reduction of postmenstrual bleeding will be measured at the 3-month and 6-month.
* Subsequent fertility outcome

ELIGIBILITY:
Inclusion Criteria:

History of cesarean section Postmenstrual and or intermenstrual spotting Large Cesarean scar niche, depth more than 50% of adjacent myometrial thickness (AMT).

Failed medical treatment Signed informed consent.

Exclusion Criteria:

A contraindication for a hysteroscopic niche resection Women with a positive pregnancy test. A contraindication for general or local anaesthesia. Coagulation disorders that lead to higher risks on bleeding or anticoagulant use.

A (suspected) malignancy, endometrial polyps, atypical endometrial cells, cervical dysplasia, hydrosalpinx that may communicate with the uterus.

Adenomyosis or leiomyoma (the International Federation of Gynecology and Obstetrics (FIGO) leiomyomia subclassification system Type 0, 1, 2, 3) or large leiomyomas causing the uterine cavity length to be ≥ 9 cm as examined by transvaginal ultrasound or MRI.

Endocrine disorders that interfere with the menstrual cycle. Irregular menstrual cycle (>35 days or intercycle variation of 2 weeks or more).

Patients who are not willing to conceive before and/or after the hysteroscopic surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
change of the residual myometrium thickness | will be measured at the 3-month and 6-month
  ultrasound measurement of the residual myometrium will be done
reduction of postmenstrual bleeding | will be assessed at the 3-month and 6-month
  participants will report their perception of the amount of bleeding using a questionnaire

SECONDARY OUTCOMES:
Subsequent fertility outcome | 1 year
  the incidence of subsequent conception following intervention will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
data may be used for another study

REFERENCES:
- [Background] Almarzuki, U. H., Ahmed, T. A. F., AlBehedy, T. M., et al. (2022). Evaluation of Anatomical Characteristics of Cesarean Scar Niche by Sonohysterography and Diagnostic Hysteroscopy in Women with Secondary Infertility. The Egyptian Journal of Hospital Medicine, 88(1), 2904-2909.
- [Background] Bakaviciute G, Spiliauskaite S, Meskauskiene A, Ramasauskaite D. Laparoscopic repair of the uterine scar defect - successful treatment of secondary infertility: a case report and literature review. Acta Med Litu. 2016;23(4):227-231. doi: 10.6001/actamedica.v23i4.3424. PMID 28356813
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Donnez O, Donnez J, Orellana R, Dolmans MM. Gynecological and obstetrical outcomes after laparoscopic repair of a cesarean scar defect in a series of 38 women. Fertil Steril. 2017 Jan;107(1):289-296.e2. doi: 10.1016/j.fertnstert.2016.09.033. Epub 2016 Nov 2. PMID 27816234
- [Background] Cohen SB, Bouaziz J, Bar On A, Orvieto R. Fertility success rates in patients with secondary infertility and symptomatic cesarean scar niche undergoing hysteroscopic niche resection. Gynecol Endocrinol. 2020 Oct;36(10):912-916. doi: 10.1080/09513590.2020.1716327. Epub 2020 Jan 27. PMID 31984814
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Stegwee SI, Beij A, de Leeuw RA, Mokkink LB, van der Voet LF, Huirne JAF. Niche-related outcomes after caesarean section and quality of life: a focus group study and review of literature. Qual Life Res. 2020 Apr;29(4):1013-1025. doi: 10.1007/s11136-019-02376-6. Epub 2019 Dec 16. PMID 31845165
- [Background] Vervoort A, Vissers J, Hehenkamp W, Brolmann H, Huirne J. The effect of laparoscopic resection of large niches in the uterine caesarean scar on symptoms, ultrasound findings and quality of life: a prospective cohort study. BJOG. 2018 Feb;125(3):317-325. doi: 10.1111/1471-0528.14822. Epub 2017 Aug 28. PMID 28703935
- [Background] Vrijdaghs V, Dewilde K, Froyman W, Van den Bosch T. Hysteroscopic management of caesarean scar defects. J Obstet Gynaecol. 2022 Jul;42(5):816-822. doi: 10.1080/01443615.2021.2003310. Epub 2022 Jan 11. PMID 35014923